CLINICAL TRIAL: NCT06345521
Title: A Comprehensive Research of Pediatric Heart Failure-- Etablishment of Follow-up System and End-Stage Heart Registration Platform for Pediatric Heart Failure
Brief Title: Etablishment of Follow-up System and End-Stage Heart Registration Platform for Pediatric Heart Failure
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Peking University First Hospital (Other); Beijing Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1-4032-3
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Congenital; End-stage Heart Failure
Keywords: Congenital Heart Failure; Registry; End-stage Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- End-Stage Heart Failure Group: Children with end-stage heart failure
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Establish a follow-up management system for pediatric heart failure and a registration platform for end-stage heart failure

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 14 years of age
* refractory heart failure

Exclusion Criteria:

-

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with end-stage heart failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-22 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of heart failure | 6 months
  During follow-up visits, echocardiographic examination is conducted to measure the left ventricular function. If LVEF falls under 55%, it is recorded as a recurrence.

SECONDARY OUTCOMES:
NT-proBNP level | 6 months
  The trend in NT-proBNP levels.
Incidence rate of drug adverse reactions | 6 months
  The incidence of abnormalities in complete blood count, electrolytes, liver and kidney function, and cardiac enzymes.
Readmission rate for heart failure | 6 months
  During follow-up visits, readmission for heart failure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No